CLINICAL TRIAL: NCT00378456
Title: Vitamins and Minerals for Children With Downs Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Child Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 98CH11
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Last update posted 2006-09-20 (Estimated); Status verified 2006-09

CONDITIONS: Trisiomy 21 (Down Syndrome)
MeSH Terms: conditions — Down Syndrome | interventions — Antioxidants; Zinc; Leucovorin

INTERVENTIONS:
Drug: Antioxidants- (Vitamins A,C,E Selenium and Zinc)
Drug: Folinic acid
Drug: Vitamins A,C,E Selenium and Zinc and Folinic acid.
Drug: Placebo

SUMMARY:
The trial aimed to examine the effects of supplementation with antioxidants and folinic acid on the health, growth and psychomotor development of children with Down syndrome. 156 children with Trisomy 21, less than 7 months of age were recruited and randomised into four groups to receive antioxidants, folinic acid, a combination of antioxidants and folinic acid or a placebo. Blinded outcome assessment was carried out 18 months later.Blood and urine samples were also taken around 12 months of age to examine metabolic effects of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Under 7 months of age
* Trisomy 21
* Live in recruitment Area-i.e. London inside M25, in West Midlands or SW England.
* One parent speaks English

Exclusion Criteria:

* No life threatening cardiac disease

Ages: 0 Years to 7 Months | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Logan, Principal Investigator — Peninsular Medical School, Exeter
Locations (3):
- United Kingdom (3):
  - Institute of Child Health, Birmingham
  - Peninsular Medical School, Exeter
  - Institute of Child Health, London, London

REFERENCES:
- [Derived] Ellis JM, Tan HK, Gilbert RE, Muller DP, Henley W, Moy R, Pumphrey R, Ani C, Davies S, Edwards V, Green H, Salt A, Logan S. Supplementation with antioxidants and folinic acid for children with Down's syndrome: randomised controlled trial. BMJ. 2008 Mar 15;336(7644):594-7. doi: 10.1136/bmj.39465.544028.AE. Epub 2008 Feb 21. PMID 18296460
- [Derived] Ellis J, Logan S, Pumphrey R, Tan HK, Henley W, Edwards V, Moy R, Gilbert R. Inequalities in provision of the Disability Living Allowance for Down syndrome. Arch Dis Child. 2008 Jan;93(1):14-6. doi: 10.1136/adc.2006.112839. Epub 2007 Mar 7. PMID 17344250